CLINICAL TRIAL: NCT03073317
Title: PREPARE, Prematurity Reduction by Pre-eclampsia Care
Acronym: PREPARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Fernandes Figueira (Other Government)
Collaborators: CoLab (Unknown); SMSDC/RJ (Unknown); University of Campinas, Brazil (Other); UPECLIN HC FM Botucatu Unesp (Other); HGA (Unknown); HOSPITAL MATERNIDADE LEONOR MENDES DE BARROS (Unknown); Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Principal Investigator, Marcos Augusto Bastos Dias, PhD, Instituto Fernandes Figueira
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: PRES-023-PPE-15
Record Dates: First submitted 2017-02-21; First posted 2017-03-08 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Pre-Eclampsia; Premature Birth
Keywords: Preterm Infants; Premature Birth; Placenta growth factor; Prenatal Care; PERINATAL MORTALITY; Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia; Premature Birth; Perinatal Death

STUDY DESIGN:
Intervention Model Description: stepped-wedge cluster-randomised trial in seven clusters
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- INTERVENTION (Experimental): Clinical protocol using FullPIERS and sFlit/PLGF ratio (Soluble fms-Like Tyrosine Kinase-1-to-Placental Growth Factor Ratio)
  Interventions: Diagnostic Test: FullPIERS and sFlit/PLGF (Soluble fms-Like Tyrosine Kinase-1-to-Placental Growth Factor Ratio)
- CONTROL (No Intervention): Usual clinic control

INTERVENTIONS:
Diagnostic Test: FullPIERS and sFlit/PLGF (Soluble fms-Like Tyrosine Kinase-1-to-Placental Growth Factor Ratio) — Once the centre is randomised to receive the intervention, all eligible women will have serum sFlt1/PlGF measurement performed and fullPIERS assessment and both results will be revealed to the care providers. This will include all women with pre-eclampsia or suspected pre-eclampsia cared for at the main hospital centres (and not be limited to women referred to the hospital from the community health centres). sFlt-1/PlGF will be tested by immunoassays (Roche Platform®). The result read out is provided by specific machines provided by Roche in less than one hour, which permits rapid clinical decision-making. Risk stratification using fullPIERS will be performed on tablet computers using a pre-defined risk scoring system integrated within the MedSciNet database.
  Arms: INTERVENTION

SUMMARY:
Investigators will test a novel system of integrated care, to promote the use of the WORLD HEALTH ORGANIZATION Guidelines for the management of pre-eclampsia and initiate the use of a structured risk assessment strategy to reduce the incidence of preterm delivery from pre-eclampsia by providing obstetricians with the confidence to safely defer delivery of women with pre-eclampsia, identified to be of low risk.

DETAILED DESCRIPTION:
This proposal (PREPARE), led by Brazilian investigators in collaboration with the Global Pregnancy Collaboration (CoLab) is centred on 7 hospital centres and their 23 satellite community health centres (UBSs). There are two clinical initiatives: First, a programme of systematic knowledge transfer (KT) to encourage adoption of the WHO Guidelines to prevent pre-eclampsia as part of routine antenatal care (Objective 1); second an intervention to reduce unnecessary preterm deliveries for the management of pre-eclampsia. CoLab investigators have developed methods to identify those women with preterm pre-eclampsia whose pregnancies can be safely prolonged.4-6 In Objective 2.1, these methods will be applied to women presenting with definite or suspected pre-eclampsia at < 37 weeks' gestation. Investigators will determine the likelihood of an imminent adverse outcome in these women using Soluble fms-Like Tyrosine Kinase-1-to-Placental Growth Factor Ratio (sFlT-1/PlGF) measurement and fullPIERS clinical assessment. Prior studies with these approaches indicate more than 98% negative predictive value for adverse outcomes for both.4-6 Investigators will delay delivery in those whose risk is low, caring for patients in accordance with evidence-based WHO guidelines.Unlike medications, management cannot be tested in a blinded way. Management needs integrated skills and commitment from caregivers. Hence, a standard randomized controlled trial is inappropriate. Instead investigators propose a Stepped Wedge Design to study outcomes in the 7 geographically diverse study centres, throughout Brazil. At least 6 women with preterm pre-eclampsia will deliver at each centre every month. The primary outcome will be a lower rate of PRETERM BIRTH due to pre-eclampsia as a proportion of total deliveries in the centre(s) after implementation of the plan compared to prior to its introduction. The study will have 80% power to demonstrate a 25% reduction (2.0 - 1.5%). Investigators will assess maternal and foetal adverse events as secondary outcomes. Objective 2.2 will institute an intense program of knowledge transfer to implement the new management techniques. In Objectives 2.3 and 2.4 will determine patient and provider satisfaction and the economic impact of the care plan. In Objective 3 will establish a biobank and database to begin to assess demographic factors and biological analytes that may help identify unique predictive and diagnostic/pathophysiological features for pre-eclampsia in the Brazilian population (that may extend to other low and middle income countries (LMIC)). For two years at routine visits (≤16 weeks, 28-32 weeks) at each UBS, relevant data and plasma, serum, urine and DNA samples will be stored to the appropriate standards in the biorepository (at least 7000 cases). Investigators estimate that will acquire samples at delivery in at least 5000 of these women. For four years, biological samples from women with pre-eclampsia or other adverse outcomes and 2 matched controls will be collected at admission for labour (an additional 3,000 subjects). Objective 4 will initiate pilot studies to identify novel biomarkers, and compare these and other known pathophysiological factors with those from LMIC (Africa, India) and HIC using samples from CoLab. Additional funding will be sought for expansion and validation (e.g. Merck for Mothers). Investigators will also seek funding to address risk stratification in apparently low risk women, based on the samples collected at 28-32 weeks. Objective 5 will promote intellectual interactions and collaboration between the seven centres and CoLab. Ability to understand and cure complex adverse pregnancy outcomes leading to acute and long-range disability in children requires intensive collaboration across usual "silos" including hospitals and nations. The coordinators anticipate the interaction of investigators and care providers in the seven centres will foster intellectual collaboration and improved standardized care. Brazilian investigators will become members of CoLab, increasing its unique vision, expertise and resources (current data and biological materials from 28 centres). worldwide).

ELIGIBILITY:
Inclusion Criteria:

* pregnancy before 16 weeks
* delivery at designed maternity center

Exclusion Criteria:

* not viable fetus

Ages: 10 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1250 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-06-20 (Actual)

PRIMARY OUTCOMES:
patients with preterm preeclampsia | researchers will be assessing and reporting outcome through month 1 to month 34 of the study
  proportion of women delivered in the centres with preterm pre-eclampsia (deliveries with preterm pre-eclampsia/ total deliveries), where preterm is <37 weeks' gestation

SECONDARY OUTCOMES:
proportion of women delivered in the centers who delivered prematurely | researchers will be assessing and reporting outcome through month 1 to month 34 of the study
  proportion of women delivered with preterm pre-eclampsia/ total deliveries for pre-eclampsia, where preterm is <37 weeks' gestation
proportion of women delivered in the centres with preterm pre-eclampsia | researchers will be assessing and reporting outcome through month 1 to month 34 of the study
  proportion of women delivered in the centres with preterm pre-eclampsia (deliveries with preterm pre-eclampsia/ total deliveries), where preterm is <34 weeks' gestation
RATE PRETERM PRE-ECLAMPSIA DELIVERIES | researchers will be assessing and reporting outcome through month 1 to month 34 of the study
  proportion of women delivered with preterm pre-eclampsia/ total deliveries for pre-eclampsia, where preterm is <34 weeks' gestation
maternal morbidity and mortality defined as a composite of maternal mortality and features of 4a-4f | researchers will be assessing and reporting outcome through month 1 to month 34 of the study
  4a. HELLP syndrome cases of HELLP syndrome in women with pre-eclampsia
  4b. pulmonary oedema cases of pulmonary oedema in women with pre-eclampsia
  4c. eclampsia proportion of women with eclampsia
  4d. cerebrovascular accident (CVA) cases of maternal cerebrovascular accident (stroke or coma) in women with pre-eclampsia
  4e. renal dysfunction cases of renal dysfunction in women with pre-eclampsia, where criteria is serum creatinine of >150
frequency of severe hypertension | researchers will be assessing and reporting outcome through month 1 to month 34 of the study
  systolic BP ≥ 160 mmHg or diastolic BP ≥ 110 mm/Hg
placental abruption | researchers will be assessing and reporting outcome through month 1 to month 34 of the study
  cases of placental abruption
mode of delivery (total C-sections) | researchers will be assessing and reporting outcome through month 1 to month 34 of the study
  total number of reported C-sections
stillbirth | researchers will be assessing and reporting outcome through month 1 to month 34 of the study
  cases of stillbirth at >20 weeks
early neonatal mortality | researchers will be assessing and reporting outcome through month 1 to month 34 of the study
  cases of neonatal mortality at <7 days
admission to the neonatal care unit | researchers will be assessing and reporting outcome through month 1 to month 34 of the study
  cases of admission to the neonatal care unit due to prematurity related to pre-eclampsia

CONTACTS AND LOCATIONS:
Overall Officials: Marcos A Dias, PhD, Principal Investigator — Instituto Fernandes Figueira
Locations (8):
- Brazil (8):
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, RIO GDE DO SUL
  - Maternidade Unesp Botucatu, Botucatu, São Paulo
  - Caism - Unicamp, Campinas, São Paulo
  - Hospital Guilherme Alvaro, Santos, São Paulo
  - Instituto Fernandes Figueira, Rio de Janeiro
  - Maternidade Maria Amelia Buarque de Holanda, Rio de Janeiro
  - Maternidade Leila Diniz, Rio de Janeiro
  - Hospital Maternidade Leonor Mendes de Barros, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ananth CV, Vintzileos AM. Medically indicated preterm birth: recognizing the importance of the problem. Clin Perinatol. 2008 Mar;35(1):53-67, viii. doi: 10.1016/j.clp.2007.11.001. PMID 18280875
- [Result] Redman CW, Sargent IL. Latest advances in understanding preeclampsia. Science. 2005 Jun 10;308(5728):1592-4. doi: 10.1126/science.1111726. PMID 15947178
- [Result] WHO Recommendations for Prevention and Treatment of Pre-Eclampsia and Eclampsia. Geneva: World Health Organization; 2011. Available from http://www.ncbi.nlm.nih.gov/books/NBK140561/ PMID 23741776
- [Result] Zeisler H, Llurba E, Chantraine F, Vatish M, Staff AC, Sennstrom M, Olovsson M, Brennecke SP, Stepan H, Allegranza D, Dilba P, Schoedl M, Hund M, Verlohren S. Predictive Value of the sFlt-1:PlGF Ratio in Women with Suspected Preeclampsia. N Engl J Med. 2016 Jan 7;374(1):13-22. doi: 10.1056/NEJMoa1414838. PMID 26735990
- [Result] von Dadelszen P, Payne B, Li J, Ansermino JM, Broughton Pipkin F, Cote AM, Douglas MJ, Gruslin A, Hutcheon JA, Joseph KS, Kyle PM, Lee T, Loughna P, Menzies JM, Merialdi M, Millman AL, Moore MP, Moutquin JM, Ouellet AB, Smith GN, Walker JJ, Walley KR, Walters BN, Widmer M, Lee SK, Russell JA, Magee LA; PIERS Study Group. Prediction of adverse maternal outcomes in pre-eclampsia: development and validation of the fullPIERS model. Lancet. 2011 Jan 15;377(9761):219-27. doi: 10.1016/S0140-6736(10)61351-7. Epub 2010 Dec 23. PMID 21185591
- [Result] Dantas EM, Pereira FV, Queiroz JW, Dantas DL, Monteiro GR, Duggal P, Azevedo Mde F, Jeronimo SM, Araujo AC. Preeclampsia is associated with increased maternal body weight in a northeastern Brazilian population. BMC Pregnancy Childbirth. 2013 Aug 8;13:159. doi: 10.1186/1471-2393-13-159. PMID 23927768
- [Result] Kajantie E, Eriksson JG, Osmond C, Thornburg K, Barker DJ. Pre-eclampsia is associated with increased risk of stroke in the adult offspring: the Helsinki birth cohort study. Stroke. 2009 Apr;40(4):1176-80. doi: 10.1161/STROKEAHA.108.538025. Epub 2009 Mar 5. PMID 19265049
- [Result] Passini R Jr, Tedesco RP, Marba ST, Cecatti JG, Guinsburg R, Martinez FE, Nomura ML; Brazilian Network of Studies on Reproductive and Perinatal Health. Brazilian multicenter study on prevalence of preterm birth and associated factors. BMC Pregnancy Childbirth. 2010 May 19;10:22. doi: 10.1186/1471-2393-10-22. PMID 20482822
- [Result] Camargo EB, Moraes LF, Souza CM, Akutsu R, Barreto JM, da Silva EM, Betran AP, Torloni MR. Survey of calcium supplementation to prevent preeclampsia: the gap between evidence and practice in Brazil. BMC Pregnancy Childbirth. 2013 Nov 11;13:206. doi: 10.1186/1471-2393-13-206. PMID 24215470
- [Result] Chappell LC, Milne F, Shennan A. Is early induction or expectant management more beneficial in women with late preterm pre-eclampsia? BMJ. 2015 Apr 10;350:h191. doi: 10.1136/bmj.h191. No abstract available. PMID 25861796
- [Result] Vigil-De Gracia P, Reyes Tejada O, Calle Minaca A, Tellez G, Chon VY, Herrarte E, Villar A, Ludmir J. Expectant management of severe preeclampsia remote from term: the MEXPRE Latin Study, a randomized, multicenter clinical trial. Am J Obstet Gynecol. 2013 Nov;209(5):425.e1-8. doi: 10.1016/j.ajog.2013.08.016. Epub 2013 Aug 14. PMID 23954534
- [Result] von Dadelszen P, Magee LA, Roberts JM. Subclassification of preeclampsia. Hypertens Pregnancy. 2003;22(2):143-8. doi: 10.1081/PRG-120021060. PMID 12908998
- [Result] Brown CA, Lilford RJ. The stepped wedge trial design: a systematic review. BMC Med Res Methodol. 2006 Nov 8;6:54. doi: 10.1186/1471-2288-6-54. PMID 17092344
- [Result] Hussey MA, Hughes JP. Design and analysis of stepped wedge cluster randomized trials. Contemp Clin Trials. 2007 Feb;28(2):182-91. doi: 10.1016/j.cct.2006.05.007. Epub 2006 Jul 7. PMID 16829207
- [Result] Harvey G, Loftus-Hills A, Rycroft-Malone J, Titchen A, Kitson A, McCormack B, Seers K. Getting evidence into practice: the role and function of facilitation. J Adv Nurs. 2002 Mar;37(6):577-88. doi: 10.1046/j.1365-2648.2002.02126.x. PMID 11879422
- [Result] von Dadelszen P, Sawchuck D, McMaster R, Douglas MJ, Lee SK, Saunders S, Liston RM, Magee LA; Translating Evidence-Based Surveillance and Treatment Strategies (TESS) Group. The active implementation of pregnancy hypertension guidelines in British Columbia. Obstet Gynecol. 2010 Sep;116(3):659-666. doi: 10.1097/AOG.0b013e3181eb669d. PMID 20733449
- [Result] Roberts JM, Hubel CA. The two stage model of preeclampsia: variations on the theme. Placenta. 2009 Mar;30 Suppl A(Suppl A):S32-7. doi: 10.1016/j.placenta.2008.11.009. Epub 2008 Dec 13. PMID 19070896
- [Result] Myers JE, Kenny LC, McCowan LM, Chan EH, Dekker GA, Poston L, Simpson NA, North RA; SCOPE consortium. Angiogenic factors combined with clinical risk factors to predict preterm pre-eclampsia in nulliparous women: a predictive test accuracy study. BJOG. 2013 Sep;120(10):1215-23. doi: 10.1111/1471-0528.12195. Epub 2013 Mar 21. PMID 23906160
- [Derived] De Oliveira L, Roberts JM, Jeyabalan A, Blount K, Redman CW, Poston L, Seed PT, Chappell LC, Dias MAB; PREPARE trial group. PREPARE: A Stepped-Wedge Cluster-Randomized Trial to Evaluate Whether Risk Stratification Can Reduce Preterm Deliveries Among Patients With Suspected or Confirmed Preterm Preeclampsia. Hypertension. 2023 Oct;80(10):2017-2028. doi: 10.1161/HYPERTENSIONAHA.122.20361. Epub 2023 Jul 11. PMID 37431663
- [Derived] Dias MAB, De Oliveira L, Jeyabalan A, Payne B, Redman CW, Magee L, Poston L, Chappell L, Seed P, von Dadelszen P, Roberts JM; PREPARE Research Group. PREPARE: protocol for a stepped wedge trial to evaluate whether a risk stratification model can reduce preterm deliveries among women with suspected or confirmed preterm pre-eclampsia. BMC Pregnancy Childbirth. 2019 Oct 7;19(1):343. doi: 10.1186/s12884-019-2445-x. PMID 31590640